CLINICAL TRIAL: NCT00167570
Title: Long Term Clinical Evaluation of SLS Transtibial Sockets
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: VA-A2755-r-UT-001-0011-267; VA-A2755-r
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2012-09

CONDITIONS: Trauma; Diabetes
Keywords: Artificial Limbs; Amputees; Computer-Aided Design
MeSH Terms: conditions — Wounds and Injuries; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Prosthetic socket fabricated using selective laser sintering

SUMMARY:
The overall long-term goal of this project is the development of a clinically practical system for rapid prosthetic limb provision that integrates computer-aided design with solid freeform fabrication techniques. This proposal builds on our previous successful demonstration of the feasibility of SFF socket fabrication and will address several key issues that underlie its clinical viability. The specific objectives of the proposed work are:

1. To develop improved designs for SFF transtibial prosthetic sockets that allow the use of industry standard pylon mounts and incorporate variable compliance elements.
2. Determine the clinical effectiveness of variable wall compliance elements in enhancing the comfort and fit of transtibial prosthetic sockets.
3. Determine the durability and functionality of SFF sockets during extended clinical use.

These objectives will be met over a three-year period. The initial phase of the proposed work will use an iterative engineering design - modeling - evaluation process to develop variable compliance elements and an industry standard pylon mount adapter. During the second phase of the proposed work, clinical evaluations of SFF prosthetic sockets will be studied. The effectiveness of variable compliant elements in enhancing comfort and fit will be determined using a within subject case comparison study of SFF sockets with conventional laminated sockets. Durability of SFF sockets that incorporate an industry standard pylon mounting system will be determined during a 12-month clinical field trial.

DETAILED DESCRIPTION:
Successful rehabilitation for the majority of lower extremity amputees includes prosthetic limb fitting and training. Critical to the success of prosthetic fitting is a comfortable, well fitting socket. Accomplishing this remains a clinical challenge with residual limb pain and socket discomfort affecting 20-55% of lower limb amputees. Achieving an acceptable socket fit using conventional prosthetic techniques requires individual custom molding and fabrication in a labor intensive, costly process. Alternative methods of fabricating prosthetic sockets that can improve efficiency in prosthetic provision, enhance comfort and fit, or reduce cost are needed to ensure the continued optimal rehabilitation of the amputee. This project will continue the development of a new promising method of socket fabrication using solid freeform fabrication (SFF) based on selective laser sintering (SLS) technology. SFF allows the direct manufacture of a prosthetic socket without the intermediate molds and laminating process required with conventional techniques.

The overall long-term goal of this project is the development of a clinically practical system for rapid prosthetic limb provision that integrates computer-aided design with solid freeform fabrication techniques. This proposal builds on our previous successful demonstration of the feasibility of SFF socket fabrication and will address several key issues that underlie its clinical viability. The specific objectives of the proposed work are:

1. To develop improved designs for SFF transtibial prosthetic sockets that allow the use of industry standard pylon mounts and incorporate variable compliance elements.
2. Determine the clinical effectiveness of variable wall compliance elements in enhancing the comfort and fit of transtibial prosthetic sockets.
3. Determine the durability and functionality of SFF sockets during extended clinical use.

These objectives will be met over a three-year period. The initial phase of the proposed work will use an iterative engineering design - modeling - evaluation process to develop variable compliance elements and an industry standard pylon mount adapter. During the second phase of the proposed work, clinical evaluations of SFF prosthetic sockets will be studied. The effectiveness of variable compliant elements in enhancing comfort and fit will be determined using a within subject case comparison study of SFF sockets with conventional laminated sockets. Durability of SFF sockets that incorporate an industry standard pylon mounting system will be determined during a 12-month clinical field trial.

ELIGIBILITY:
Inclusion Criteria:

All subjects will be lower extremity amputees of at least one year duration and are 18 years of age or older.

They must meet the Medicare Functional Classification Level K2 or K3 class for prosthetic use (unlimited household or limited community level ambulator).

Exclusion Criteria:

There must be no current stump wounds or breakdown or a history of repeated skin breakdown with adequately fitting prostheses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2003-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Durability during household and community mobility. | Up to 12 months
  Subjects were followed for up to 12 months in 3 months intervals for examination of the physical condition of socket and for subject gait assessment with socket

SECONDARY OUTCOMES:
User perceptions of comfort, fit, and function. | Up to 12 months
  Subjects were followed up at 3 month intervals and assessed for comfort fit and function

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Walsh, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- South Texas Veterans Healthcare System, San Antonio, Texas, United States